CLINICAL TRIAL: NCT05398042
Title: Effect of Oral Ketone Administration During Inactivity-induced Muscle Atrophy and Retraining-induced Regeneration
Brief Title: Ketone Administration During Inactivity and Retraining
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Peter Hespel, Principal Investigator, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S65695
Record Dates: First submitted 2021-12-06; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Exercise; Healthy Male/Female Subjects
Keywords: Ketone; Inactivity-induced muscle atrophy; Retraining-induced regeneration
MeSH Terms: conditions — Motor Activity; Ketosis | interventions — formic acid 4-(3-oxobutyl)phenyl ester; Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Ketone placebo will be provided
  Interventions: Dietary Supplement: Medium Chain Triglyceride (MCT) oil
- Ketone (Experimental): Ketone esters will be provided
  Interventions: Dietary Supplement: Ketone ester

INTERVENTIONS:
Dietary Supplement: Ketone ester — A daily dose of 3x20g of ketone ester supplementation during a six week intervention period
  Arms: Ketone
Dietary Supplement: Medium Chain Triglyceride (MCT) oil — A daily dose of 3x12.8g of MCT oil supplementation during a six week intervention period
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate the effect of oral ketone administration during inactivity-induced muscle atrophy and retraining-induced regeneration. Potential changes in muscle function (cycling performance, knee-extension force and power, jump height) and mass, blood flow and the muscular extracellular matrix will be the main focus. In this context, the dominant leg of the participants (n=24) will be immobilized with a brace for 2 weeks and subsequently retrained in a 4-week progressive resistance exercise training program to stimulate muscle regeneration. During the immobilization and rehabilitation period, participants receive either ketone ester (KE) or placebo (CON). 4 experimental sessions are performed during this time frame in order to evaluate the effects of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Recreational sports participation, including general fitness training, between 2 and 5 hours max per week
* Good health status confirmed by a medical screening
* Body mass index between 18 and 25

Exclusion Criteria:

* Any kind of injury/pathology that is a contra-indication to perform resistance exercise
* Intake of any medication or nutritional supplement that could impact muscle protein synthesis during the period of the study
* Intake of any whey protein, casein or branched-chain amino acid supplement or anti-inflammatory drug from 1 month prior to the start of the study
* Blood donation within 3 months prior to the start of the study
* Smoking
* Pregnant
* More than 3 alcoholic beverages per day
* Current participation in another research trial
* Any other argument to believe that the subject is unlikely to successfully complete the full study protocol
* Adherence to a high-fat, low-carbohydrate ketogenic diet (less than 20% of energy intake derived from carbohydrates)
* (Cow's) milk protein allergy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-06-20 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Exercise performance | Day 0 - day 14 - day 28 - day 42
  Changes in exercise performance as evaluated during a graded exercise test
Echo-Doppler measurement of femoral artery | Day 0 - Day 14 - Day 28 - Day 42
  Change in blood flow of arteria femoralis
Muscle volume | Day 0 - Day 14 - Day 28 - Day 42
  Change in volume of quadriceps evaluated by computed-tomography scan
Muscular functional capacity | Day 0 - Day 14 - Day 28 - Day 42
  Change in mean power produced during 30 unilateral knee extensions on a knee-extension apparatus
Skeletal muscle biopsies | Day 0 - Day 14 - Day 28 - Day 42
  Changes in myofibrillar protein synthesis
Skeletal muscle biopsies | Day 0 - Day 14 - Day 28 - Day 42
  Changes in connective tissue protein synthesis
Blood marker of collagen synthesis | Day 0 - Day 14 - Day 28 - Day 42
  Change in PINP (n-terminal peptide of pro-collagen I) concentration in blood

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Physiology Research Group, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided